CLINICAL TRIAL: NCT03399097
Title: Characterizing the Intestinal Hormonal Secretion in Non-obese, Obese and Non-obese Patients After Bariatric Surgery
Status: Withdrawn | Type: Observational
Why Stopped: change sites
Sponsor: Dr. Ofir Harnoy MD (Other Government)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor-Investigator, Dr. Ofir Harnoy MD, Principal Investigator, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Other Study IDs: 3830-17-SMC
Record Dates: First submitted 2017-12-20; First posted 2018-01-16 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-obese: non-obese
- obese: obese
- previously obese: previously obese

SUMMARY:
The enteroendocrine system is composed from different cells along the different parts of the gastrointestinal tract, secreting diverse hormones and bariatric surgery alters intestinal hormone secretion, affecting glycemic control and weight. The aim of the study is to characterize the composition and secretory profile of enteroendocrine cells in the obese, non-obese and non-obese post bariatric surgery.

DETAILED DESCRIPTION:
Obesity and Diabetes Mellitus (DM) impose a significant burden of morbidity on many individuals around the world. In recent years, the enteroendocrine cells system with its diverse hormones (Glucagon, GLP-1, GIP and others) was increasingly recognized as a key player in obesity and DM homeostasis.

Bariatric surgery induces weight loss as well as an improvement in glycemic control often leading to diabetes reversal and occasionally to postprandial hypoglycemic events. The aim of the study is to characterize the composition and secretory profile of enteroendocrine cells in the obese, non-obese and non-obese post bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* BMI>= 35 or BMI<=25 or 6-12 months after RYGB surgery

Exclusion Criteria:

* Known HIV infection
* Any NSAID'S usage in the last 3 months
* Known Celiac disease
* Concomitant disease with potential small bowel or colonic involvement (Tb, sarcoidosis, IBD, microscopic colitis etc')
* Pregnancy
* Participation in another clinical trial
* Any use of medications known to modulate glucagon levels such as GLP1 analogs, DPP4 inhibitors and/or SGLT2 inhibitors.
* Insulin-treated patients.
* Declined to sign an informed consent

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that are referred for screening colonoscopy in the gastroenterology department.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Characterization the composition of enteroendocrine cells in the obese, non-obese and non-obese post-bariatric surgery. | 3 years
  The number of somatostatin, proglucagon and serotonin positive cells in the terminal ileum and Colon by immunohistochemistry.

SECONDARY OUTCOMES:
Characterization the secretory profile of enteroendocrine cells in the obese, non-obese and non-obese post-bariatric surgery. | 4 YEARS.
  Total hormonal content of somatostatin, proglucagon and serotonin will be quantified using mRNA level qunatitation

OTHER OUTCOMES:
Characterization the secretory profile of enteroendocrine cells in the obese, non-obese and non-obese post-bariatric surgery. | 4 years
  Total hormonal content of somatostatin, proglucagon and serotonin will be quantified using ELISA.
Characterization the location of enteroendocrine cells in the obese, non-obese and non-obese post-bariatric surgery. | 4 years.
  The location of somatostatin, proglucagon and serotonin will be quantified using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Tirosh, MD, PhD, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel